CLINICAL TRIAL: NCT02363426
Title: Randomized Controlled Open-Label Non-Inferiority Trial Comparing Day 5 Embryos Derived From Intravaginal Culture Using the Medical Device INVOcell to Traditional In Vitro Fertilization
Brief Title: Vaginal Culture Using INVOcell Compared to Traditional IVF Incubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Invaron Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-006
Record Dates: First submitted 2015-02-05; First posted 2015-02-16 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: intravaginal culture; in vitro fertilization; blastocyst; pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Device: INVOcell Culture Device (Other): 5 day oocyte incubation using INVOcell Culture Device within the vaginal cavity.
  Interventions: Device: INVOcell Culture Device
- Medical Device: IVF Incubator (Active Comparator): 5 day oocyte incubation using traditional IVF incubation.
  Interventions: Device: IVF Incubation

INTERVENTIONS:
Device: INVOcell Culture Device — INVOcell is a vaginal culture device
  Other Names: INVOcell, INVOcell Culture Device
  Arms: Medical Device: INVOcell Culture Device
Device: IVF Incubation — IVF Incubator
  Arms: Medical Device: IVF Incubator

SUMMARY:
The purpose of this study is to evaluate intravaginal culture using the medical device INVOcell to generate day 5 blastocysts in comparison to traditional IVF.

DETAILED DESCRIPTION:
This is a Phase III, single center, open label randomized comparative trial to evaluate intravaginal culture using INVOcell vs. traditional IVF to generate day 5 embryos Pilot: 40 couples (80 patients), randomized to receive either intravaginal culture (n=20) using the INVOcell or traditional IVF (n=20) Primary Endpoints: Blastocyst generation rate: number of day 5 embryos of "good quality" defined as 2BB or greater (expansion of embryo 2,3,4,5 or 6 and inner cell mass and outer cell mass grades of A or B) or higher using the Gardner Grading System divided by the number of eggs incubated Patient acceptability of INVOcell and intravaginal culture.

Secondary Endpoints: Live birth rate: number of cycles with a live birth divided by the number of cycles with embryo transfers.

Clinical pregnancy rate: number of cycles with fetal heartbeat at week 7 divided by the number of cycles with embryo transfers.

Fertilization rate: Number of embryos obtained after incubation divided by the number of oocytes placed in the device.

Embryo transfer rate: Number of cycles initiated divided by the number of cycles with embryo transfers Miscarriage rate: Number of miscarriages divided by the number of cycles with embryo transfers Multiple rate: Number cycles with twins or triplets divided by the number of cycles with embryo transfers Miscarriage rate per clinical pregnancy: Number of miscarriages divided by the number of cycles with clinical pregnancy

ELIGIBILITY:
Inclusion Criteria:

Couples who will participate to the study will be pre selected for the following major indications:

Women diagnosed with:

* Tubal factor
* Endometriosis (type I to II)
* Ovulatory dysfunction (slight)
* Multiple female factors (<2)

Males with slight male factor

Couples with:

* Unknown factor
* Multiple factors, from female and male origin (<2)
* Other rare factors not excluded by the inclusion/exclusion criteria (e.g. cervical mucus immune factor not treatable by IUI)

The pre-selected couples will be included in the study only if they fulfill the more specific inclusion and exclusion criteria below.

Couples may be included in the study only if they have been informed about the study and have given their written consent.

Infertile couple with failure to conceive a recognized pregnancy after one year (or 12 menstrual cycles) of unprotected intercourse IVF has been determined by the physician to be their next treatment

Women included in the study should:

* Be between the age of 18 and 38 (up to 38th birthday at the time of the enrollment).
* Have had a normal gynecological examination and Pap smear in the last 12 months.
* Have a normal follicle stimulating hormone (<10 mIU/mL) and E2 (<250 pmol/L) on Day 3, determined in the past 12 months
* Have an anti-mullerian hormone >1 or <3 ng/mL
* Have had a normal baseline pelvic ultrasound examination in the past 12 months
* Have a normal uterine cavity as assessed in the past year by hysterosalpingogram, sonohysterography or hysteroscopy. Prior tubal ligation is acceptable.
* Have had negative cervical tests for G.C and Chlamydia in the past 12 months. Have male partner with a normal semen analysis with a total number of > 15 million total motile spermatozoa with normal morphology or borderline normal morphology (> 3% with the strict criteria) and a progression rating of >2.

Exclusion Criteria:

Women to be excluded from this study are those who have:

* Inability to read and speak English fluently
* A history of recurrent vaginitis
* A history of toxic shock syndrome
* Known allergies to plastic, human serum proteins or gentamicin
* Had pelvic surgery within the past 8 weeks, excluding diagnostic laparoscopy
* Pelvic inflammatory disease (PID) within the past 3 months and were treated with antibiotics
* Severe endometriosis (stage III-IV) or endometriomas (past or present)
* Clinical signs of vaginal infection
* Significant abnormalities of the vaginal cavity
* Sub mucus or intramural fibroids (>1 cm diameter)
* Hydrosalpinx
* Chronic illness, e.g. autoimmune disease, diabetes
* BMI >36
* Donor oocytes, donor sperm
* antral follicle count < 6 or > 20
* Anti-Mullerian Hormone <1 or >3
* Previously responded poorly to ovarian stimulation and polycystic ovary patients
* High responder to ovarian stimulation
* Cervical stenosis, as demonstrated by failed mock embryo transfer
* Cannot tolerate a speculum examination
* Unwilling or unable to wear a retention system (diaphragm) during the 5 days of incubation.

> 2 previously failed IVF (neg βhCG)

* Previously failed fertilization of all oocytes previous IVF cycle
* Smoke or abuse drugs and alcohol
* Poor understanding of the procedure
* Partner with vasectomy reversal
* Partner with difficulty in producing sperm specimen
* Partner with uro-genital infection. Sperm culture will be performed if the partner shows or has shown some symptoms of uro-genital infection.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Blastocyst Quality | Measures assessed following 5 days incubation, approximately 17 days following randomization
  Blastocyst generation rate: number of day 5 embryos of "good quality" defined as 2BB or greater (expansion of embryo 2,3,4,5 or 6 and inner cell mass and outer cell mass grades of A or B) or higher using the Gardner Grading System divided by the number of eggs incubated

SECONDARY OUTCOMES:
Patient Acceptability | Measures assessed at first followup visit following embryo transfer, approximately 9 weeks post randomization
  Patient acceptability of INVOcell and intravaginal culture using a 12 point subjective and quantitative questionnaire.
Live Birth Rate | Measures assessed 9 months post embryo transfer, approximately 9 months and two weeks following randomization
  Live birth rate: number of cycles with a live birth divided by the number of cycles with embryo transfers.
Clinical Pregnancy Rate | Measures assessed approximately 16 days following embryo transfer, approximately 4 weeks following randomization.
  Clinical pregnancy rate: number of cycles with fetal heartbeat at week 7 divided by the number of cycles with embryo transfers.
Fertilization Rate | Measures assessed following 5 days post incubation, approximately 2 and 1/2 weeks post randomization.
  Fertilization rate: Number of embryos obtained after incubation divided by the number of oocytes placed in the device.
Embryo Transfer Rate | Measures assessed following 5 days incubation, approximately 2 and 1/2 weeks following randomization.
  Embryo transfer rate: Number of cycles initiated divided by the number of cycles with embryo transfers
Miscarriage Rate | Measures assessed following embryo transfer and a maximum of 9 months gestation.
  Miscarriage rate: Number of miscarriages divided by the number of cycles with embryo transfers
Multiple Rate | Measures assessed 9 months after the last subject received an embryo transfer, once all live birth data is known for each embryo.
  Multiple rate: Number cycles with twins or triplets divided by the number of cycles with embryo transfers

CONTACTS AND LOCATIONS:
Locations (1):
- C.A.R.E., Beford, Texas, United States

REFERENCES:
- [Background] Ranoux C, Aubriot FX, Dubuisson JB, Cardone V, Foulot H, Poirot C, Chevallier O. A new in vitro fertilization technique: intravaginal culture. Fertil Steril. 1988 Apr;49(4):654-7. doi: 10.1016/s0015-0282(16)59835-5. PMID 3350160